CLINICAL TRIAL: NCT06773403
Title: A 24 Week, Open-Label Study to Evaluate the Efficacy and Safety of Upadacitinib in Patients With Moderate-to-Severe Prurigo Nodularis
Brief Title: Upadacitinib for Prurigo Nodularis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Psoriasis Treatment Center of Central New Jersey (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETC03
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Prurigo Nodularis
MeSH Terms: interventions — upadacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Upadacitinib (Other): Open-label use of 15mg upadacitinib. Subjects have the option to increase to 30mg at week 8 if the investigator deems it necessary.
  Interventions: Drug: Upadacitinib

INTERVENTIONS:
Drug: Upadacitinib — All subject start on 15mg. At week 8 subjects may increase to 30mg if the investigators deems it necessary.

SUMMARY:
A single center, open-label study of 25 subjects to assess 24 weeks upadacitinib in patients with moderate-to-severe prurigo nodularis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult 18-64 years of age at time of screening.
2. Diagnosis of prurigo nodularis for ≥ 3 months.
3. Moderate-to-Severe prurigo nodularis as determined by at least 10 PN lesions on legs and/or arms and/or trunk at screening and baseline .
4. Failure of at least a 2-week course of medium to super potent TCS or TCS is not medically advisable for subject.
5. Females of childbearing potential must not have a positive serum pregnancy test at the Screening Visit and must have a negative urine pregnancy test at the Baseline Visit prior to study drug dosing. Note: subjects with borderline pregnancy test at Screening must have a serum pregnancy test ≥ 3 days later to determine eligibility.

   If female, subject must be postmenopausal OR permanently surgically sterile OR for females of childbearing potential practicing at least one protocol specified method of birth control, that is effective from the Baseline Visit through at least 30 days after the last dose of study drug. Female subject must not be pregnant, breastfeeding or considering becoming pregnant during the study or for approximately 30 days after the last dose of the study drug.
6. Subject is a candidate for systemic therapy per investigator discretion.
7. Able and willing to give written informed consent prior to performance of any study-related procedures.
8. Subject must be in general good health as judged by the Investigator, based on medical history, physical examination.

Exclusion Criteria:

1. Presence of skin condition other than prurigo nodularis or atopic dermatitis that may interfere with study assessments.
2. Diagnosis of active atopic dermatitis at screening and baseline.
3. PN secondary to medications.
4. PN secondary to medical conditions such as neuropathy or psychiatric disease.
5. Severe concomitant illness(es) under poor control that, in the investigator's judgment, would adversely affect the patient's participation in the study.
6. Severe renal conditions (eg, patients with uremia and/or on dialysis)
7. Participants with uncontrolled thyroid disease.
8. Active tuberculosis or non-tuberculous mycobacterial infection, or a history of incompletely treated tuberculosis unless documented adequately treated. Patients with latent TB at screening may be enrolled if tuberculosis treatment is initiated prior to first dose.
9. Diagnosed active endoparasitic infections; suspected or high risk of endoparasitic infection, unless clinical and (if necessary) laboratory assessment have ruled out active infection before randomization.
10. Active chronic or acute infection (except HIV infection) requiring treatment with systemic antibiotics, antivirals, antiprotozoals, or antifungals within 2 weeks before the screening visit or during the screening period.
11. Known or suspected immunodeficiency.
12. Active malignancy or history of malignancy within 5 years before the baseline visit, except completely treated in situ carcinoma of the cervix, completely treated and resolved non-metastatic squamous or basal cell carcinoma of the skin.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in worst-itch numeric rating scale (WI-NRS) at week 12 | 12 weeks
  Proportion of participants with improvement (change) in worst-itch numeric rating scale (WI-NRS) by ≥4 points from baseline to Week 12.

CONTACTS AND LOCATIONS:
Locations (1):
- Eczema Treatment Center of New Jersey, East Windsor, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT06773403/Prot_SAP_000.pdf